CLINICAL TRIAL: NCT04942444
Title: Dry Needling in Patients With Fibromyalgia: Analysis of Its Therapeutic Effectiveness
Brief Title: Effectiveness of Dry Needling in Fibromyalgia Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CEU San Pablo University (Other)
Responsible Party: Principal Investigator, Paula Rivas Calvo, Prof. Colaborador Doctor Paula Rivas Calvo, CEU San Pablo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEU-0021
Record Dates: First submitted 2021-02-21; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Fibromyalgia; Chronic Pain; Anxiety; Depression; Fatigue; Sleep Disorder
Keywords: dry needing
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Anxiety Disorders; Depression; Fatigue; Sleep Wake Disorders | interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients from the control group kept on taking the same medical treatment that they received before randomization
- Dry needling group (Experimental): Besides maintaining their current medical treatment, patients from the experimental group received an additional weekly one-hour session of dry needling over the 18 tender points for a 6-week-period.
  Interventions: Other: Dry needling

INTERVENTIONS:
Other: Dry needling — One-hour weekly session of DN in the 18th tender points during 6 weeks in the DNG, apart from continuing their medical treatment. The CG continue with the habitual medical treatment.
  Arms: Dry needling group

SUMMARY:
Patients with fibromyalgia (FM) complain of widespread chronic pain from deep tissues including muscles. Previous research highlights the relevance of impulse input from deep tissues for clinical FM pain. Deep dry needle stimulation is an invasive treatment modality used in the management of musculoskeletal pain. Its efficacy has been confirmed in the management of myofascial trigger points, so the purpose of the study is to determine if blocking abnormal impulse input with deep dry needling stimulation of tender point may decrease hyperalgesia, clinical pain and associated symptoms such as anxiety, depression, fatigue and improve the quality of life in FM patients.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is characterized by chronic widespread musculoskeletal pain that is often associated to other manifestations such as fatigue, sleep disturbances, anxiety and depression. FM diagnosis may be performed following the 1990 American College of Rheumatology (ACR) classification criteria that require a history of widespread pain for at least 3 months and tenderness in at least 11 of 18 defined tender points.

Dry needling is a broad term used to differentiate "non-injection" needling from the practice of "injection needling". In contrast to injection of an agent, dry needling utilizes a solid filament needle, as is used in the practice of acupuncture, and relies on the stimulation of specific reactions in the target tissue for its therapeutic effect. Is a relatively new treatment modality used by physicians and physical therapists worldwide as a part of complex treatment of chronic musculoskeletal pain. It is minimally invasive, cheap, easy to learn, and carries a low risk of complications. Its efficacy has been confirmed in numerous studies and systematic reviews on management of myofascial trigger points, acute and chronic low back pain, chronic lumbar myofascial trigger points, lumbar myofascial pain, chronic whiplash, and myofascial pain and headaches.

The clinical picture of FM suggests an increased activity and/or hypersensitivity in nociceptive pathways or inadequate activity in endogenous pain attenuation mechanisms. Administration of local injections of lidocaine in the tender points is considered a therapeutic approach in the management of FM and this therapy increases plasma concentrations of met-enkephalin. FM patients treated with dry needling also experience a rapid increase of plasma levels of met-enkephalin. Results derived from randomized clinical trials and systematic reviews disclosed no differences between injections of different substances and dry needling in the treatment of myofascial trigger points symptoms. These findings suggest that needling techniques may be effective in the management of FM.

Taken together all these considerations, the primary aim of this study is to investigate the efficacy of dry needling as a complementary treatment of severely affected FM patients. In addition, the investigators, aimed to establish whether this procedure might still yield some clinical improvement 6 weeks after the discontinuation of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had not responded to any of the previously used pharmacological and non-pharmacological treatments.
* Literate and able to complete the questionnaires and scales used in the study.
* Patients who accepted their inclusion in the trial signed the corresponding informed consent and were given an explanatory sheet of the project.

Exclusion Criteria:

* Patients with CNS involvement with or without treatment (stroke, Parkinson's, dementia, multiple sclerosis, etc.).
* Patients with inflammatory or autoimmune disease associated with Fibromyalgia.
* Patients with infectious, neoplastic disease, or parenteral drug use.
* Patients with insurmountable fear of needles
* Under 18 years of age
* Coagulation problems (including treatment with anticoagulants, due to the risk of bleeding).
* Immunosuppressed people (due to the risk of infection),
* Lymphadenectomized people (due to the risk of lymphedema)
* Hypothyroidism (due to the risk of myxedema)
* Pregnant patients
* Patients with areas of the skin that present some type of wound, infection, macula or tattoo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-01-10 (Actual); Primary Completion 2011-02-01 (Actual); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the score of pain. | -At the start of the treatment (week 0) -At the end of the 6-week intervention period (this time considered as end of intervention). -Finally, patients were again evaluated 6 week later (at week 12 after finishing the dry needling intervention)
  - Dolorimeter for assessing the myalgic score. Rank values 0 (best outcome) to 10 (worst outcome)
Changes in pain in using questionnaires | -At the start of the treatment (week 0) -At the end of the 6-week intervention period (this time considered as end of intervention). -Finally, patients were again evaluated 6 week later (at week 12 after finishing the dry needling intervention)
  Fibromyalgia Impact Questionnaire (FIQ). Rank values from 0 (best outcome) to 100 (worst outcome)
Changes in the score of pain. | At the start of the treatment (week 0) -At the end of the 6-week intervention period (this time considered as end of intervention). -Finally, patients were again evaluated 6 week later (at week 12 after finishing the dry needling intervention)
  - Visual Analogue Scale (VAS). Rank values 0 (best outcome) to 10 (worst outcome)
Changes in pain in using questionnaires | At the start of the treatment (week 0) -At the end of the 6-week intervention period (this time considered as end of intervention). -Finally, patients were again evaluated 6 week later (at week 12 after finishing the dry needling intervention)
  McGill Pain Questionnaire (MPQ) The Pain Rating Index (PRI) score indices range from 0-78 based on the rank values of the chosen words. The value (score) associated with each descriptor is based on its position or rank order in the set of words, so that the first word receives a value of 1, the next a value of 2, and so on. Range values are summed within each subclass as well as in general. The PPI (Present pain intensity) ranges from 0-5. Scoring example: Temporal Group I: Periodic (1 point), Repetitive (2 points), Insistent (3 points), Endless (4 points). Each aspect that is assessed fits into four subscales: 1 to 10, sensitive subscale, 11 to 15, affective subscale; 16, evaluative subscale; 17 to 20, subscale of diverse aspects. Especially aimed at chronic pain.
  Chronic Pain Acceptance Questionnaire (CPAQ)
Changes in pain in using questionnaires | At the start of the treatment (week 0) -At the end of the 6-week intervention period (this time considered as end of intervention). -Finally, patients were again evaluated 6 week later (at week 12 after finishing the dry needling intervention)
  Chronic Pain Acceptance Questionnaire (CPAQ). Rank values from 0 (worst outcome) to 120 (best outcome)
Changes in pain in using questionnaires | At the start of the treatment (week 0) -At the end of the 6-week intervention period (this time considered as end of intervention). -Finally, patients were again evaluated 6 week later (at week 12 after finishing the dry needling intervention)
  Pain Catastrophizing Scale (PCS). Rank values from 0 (best outcome) to 52 (worst outcome)

SECONDARY OUTCOMES:
Changes in fatigue | -At the start of the treatment (week 0) -At the end of the 6-week intervention period (this time considered as end of intervention). -Finally, patients were again evaluated 6 week later (at week 12 after finishing the dry needling intervention)
  - Six-minute walk test for the fatigue.
Changes in fatigue | -At the start of the treatment (week 0) -At the end of the 6-week intervention period (this time considered as end of intervention). -Finally, patients were again evaluated 6 week later (at week 12 after finishing the dry needling intervention)
  Visual Analogue Scale of Fatigue (VAS). Rank value from 0 (best outcome) to 10 (worst outcome)
Changes in fatigue | -At the start of the treatment (week 0) -At the end of the 6-week intervention period (this time considered as end of intervention). -Finally, patients were again evaluated 6 week later (at week 12 after finishing the dry needling intervention)
  Fatigue Severity Scale Questionnaire (FSS). Rank values from 0 (best outcome) to 63 (worst outcome)
Changes in anxiety | At the start of the treatment (week 0) -At the end of the 6-week intervention period (this time considered as end of intervention). -Finally, patients were again evaluated 6 week later (at week 12 after finishing the dry needling intervention)
  -Beck Anxiety Inventory (BAI). Rank values from 0 (best outcome) to 63 (worst outcome).
Changes in anxiety | At the start of the treatment (week 0) -At the end of the 6-week intervention period (this time considered as end of intervention). -Finally, patients were again evaluated 6 week later (at week 12 after finishing the dry needling intervention)
  - Visual Analogue Scale of Anxiety (VAS).Rank values from 0 (best outcome) to 10 (worst outcome)
Changes in Depression | At the start of the treatment (week 0) -At the end of the 6-week intervention period (this time considered as end of intervention). -Finally, patients were again evaluated 6 week later (at week 12 after finishing the dry needling intervention)
  - Beck Depression Inventory (BDI). Rank values from 0 (best outcome) to 63 (worst outcome).
Changes in Sleep | At the start of the treatment (week 0) -At the end of the 6-week intervention period (this time considered as end of intervention). -Finally, patients were again evaluated 6 week later (at week 12 after finishing the dry needling intervention)
  Pittsburgh Sleep Quality Index (PSQI). Rank values from 0 (best outcome) to 21 (worst outcome)
Changes in Quality of Life | At the start of the treatment (week 0) -At the end of the 6-week intervention period (this time considered as end of intervention). -Finally, patients were again evaluated 6 week later (at week 12 after finishing the dry needling intervention)
  * Stanford Health Assessment Questionnaire (SHAQ). Rank values from 0 (best outcome) to 3 (worst outcome).
  * Medical Outcomes Survey Short Form-36 (SF-36)
Changes in Quality of Life | At the start of the treatment (week 0) -At the end of the 6-week intervention period (this time considered as end of intervention). -Finally, patients were again evaluated 6 week later (at week 12 after finishing the dry needling intervention)
  - Medical Outcomes Survey Short Form-36 (SF-36). Rank values from 0 (worst outcome) to 100 (best outcome)

OTHER OUTCOMES:
Baseline measurements. Demographic variables. | Baseline measurements were performed after eligibility (at week 0)
  - Material status
Baseline measurements. Demographic variables. | Baseline measurements were performed after eligibility (at week 0)
  - Employment status
Baseline measurements. Demographic variables. | Baseline measurements were performed after eligibility (at week 0)
  - Education status
Baseline measurements. Demographic variables. | Baseline measurements were performed after eligibility (at week 0)
  Years until disease diagnosis
Baseline measurements. Demographic variables. | Baseline measurements were performed after eligibility (at week 0)
  - Body mass index
Baseline measurements. Demographic variables. | Baseline measurements were performed after eligibility (at week 0)
  - Number of physical symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Paula Rivas, Segovia, ESSG, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Kalichman L, Vulfsons S. Dry needling in the management of musculoskeletal pain. J Am Board Fam Med. 2010 Sep-Oct;23(5):640-6. doi: 10.3122/jabfm.2010.05.090296. PMID 20823359
- [Background] Tough EA, White AR, Cummings TM, Richards SH, Campbell JL. Acupuncture and dry needling in the management of myofascial trigger point pain: a systematic review and meta-analysis of randomised controlled trials. Eur J Pain. 2009 Jan;13(1):3-10. doi: 10.1016/j.ejpain.2008.02.006. Epub 2008 Apr 18. PMID 18395479
- [Background] Ceccherelli F, Rigoni MT, Gagliardi G, Ruzzante L. Comparison of superficial and deep acupuncture in the treatment of lumbar myofascial pain: a double-blind randomized controlled study. Clin J Pain. 2002 May-Jun;18(3):149-53. doi: 10.1097/00002508-200205000-00003. PMID 12048416
- [Background] Baldry P. Superficial versus deep dry needling. Acupunct Med. 2002 Aug;20(2-3):78-81. doi: 10.1136/aim.20.2-3.78. PMID 12216605
- [Background] Hong CZ, Hsueh TC. Difference in pain relief after trigger point injections in myofascial pain patients with and without fibromyalgia. Arch Phys Med Rehabil. 1996 Nov;77(11):1161-6. doi: 10.1016/s0003-9993(96)90141-0. PMID 8931529
- [Background] Staud R. Is it all central sensitization? Role of peripheral tissue nociception in chronic musculoskeletal pain. Curr Rheumatol Rep. 2010 Dec;12(6):448-54. doi: 10.1007/s11926-010-0134-x. PMID 20882373
- [Background] Srbely JZ, Dickey JP, Lee D, Lowerison M. Dry needle stimulation of myofascial trigger points evokes segmental anti-nociceptive effects. J Rehabil Med. 2010 May;42(5):463-8. doi: 10.2340/16501977-0535. PMID 20544158
- [Background] Wallace DJ, Linker-Israeli M, Hallegua D, Silverman S, Silver D, Weisman MH. Cytokines play an aetiopathogenetic role in fibromyalgia: a hypothesis and pilot study. Rheumatology (Oxford). 2001 Jul;40(7):743-9. doi: 10.1093/rheumatology/40.7.743. PMID 11477278